CLINICAL TRIAL: NCT05560659
Title: Lu-PSMA for Oligometastatic Prostate Cancer Treated With STereotactic Ablative Radiotherapy, a Randomised Phase II Parallel Cohort Trial
Brief Title: Lu-PSMA for Oligometastatic Prostate Cancer Treated With STereotactic Ablative Radiotherapy
Acronym: POPSTAR II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/033
Record Dates: First submitted 2022-02-17; First posted 2022-09-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Oligometastatic Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic ablative body radiotherapy (SABR) alone (No Intervention): 1-3 fractions of SABR to all sites of disease
- SABR plus 2 cycles of 177Lu-PSMA (Experimental): cycles of 177Lu-PSMA with 1-3 fractions of SABR to all sites of disease between cycle 1 and 2
  Interventions: Drug: 177Lu-PSMA

INTERVENTIONS:
Drug: 177Lu-PSMA — Lutetium-177 (177Lu)-PSMA is a radiopharmaceutical comprised of a small molecule inhibitor of PSMA that binds with high affinity to PSMA, labelled with 177Lu. 177Lu has favourable characteristics for radionuclide therapy emitting both a short-range (1-2mm) cytotoxic beta-particle, minimising irradiation of non-targeted normal tissues, alongside gamma emission that allows imaging. Numerous retrospective series initially demonstrated high clinical activity and limited normal tissue toxicity using PSMA-617 and PSMA-I&T, which are the most advanced small molecule inhibitors of PSMA, radiolabelled with 177Lu
  Arms: SABR plus 2 cycles of 177Lu-PSMA

SUMMARY:
The aim of this study is to assess the progression free survival (PFS) of SABR alone and SABR + 177Lu-prostate-specific membrane antigen (PSMA) in patients with oligometastatic prostate cancer undergoing PSMA positron emission tomography (PET) staging.

DETAILED DESCRIPTION:
Metastatic disease in patients involves treatment including systemic chemotherapy, hormonal therapy and androgen deprivation therapy. "Oligometastases" was termed to describe a state of metastatic transition wherein the cancer cells travel from the original site of tumour to other parts of the body and form fewer number of tumours. Sustained systemic therapies such as chemotherapy have been used as the Standard of care (SOC) in most cases. Novel radiotherapy like Lutetium-177 PSMA radionuclide therapy have been explored in earlier disease settings to further improve outcomes. Based on evidence from few previous trials and emerging safety data from ongoing trials, it is an effective addition to SOC to further improve patient outcomes.

The detection of prostate cancer can be done by a highly sensitive and specific test using the PSMA-PET small molecules. The evidence of high uptake of these PSMA-PET small molecules assists in selection of patients potentially suitable for novel PSMA targeted radionuclide therapy. Previous studies have demonstrated novel molecular imaging techniques, particularly PSMA PET/CT in the biochemical recurrence setting is leading to an increasing number of patients being diagnosed with oligometastatic disease which would not have been detected using conventional imaging techniques.

The Stereotactic ablative body radiotherapy (SABR) is also an emerging localised treatment option for oligometastatic prostate cancer. It delivers a highly focused beam of external radiation concentrated over a tumour and has been used to treat low volume metastatic disease to delay the use of systemic therapies. Results from previous studies show that it a safe, well-tolerated and progressively used in real-world clinical practice to treat patients with low volume of metastatic cancer. Based on the results of a previous trial done by this team, patients with one to three sites of disease treated with a single session of SABR showed promising outcomes.

The aim of this trial is to evaluate the progression free survival of SABR alone and SABR + 177Lu-prostate-specific membrane antigen (PSMA) in patients with oligometastatic prostate cancer undergoing PSMA positron emission tomography (PET) staging.

92 men with oligometastatic prostate cancer will be enrolled in this trial and split into 1:1 ratio to either stereotactic ablative body radiotherapy (SABR) alone or SABR plus 2 cycles of 177Lu-PSMA over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 years or older at screening
2. Patient has provided written informed consent
3. Histologically confirmed prostate adenocarcinoma w
4. Prior definitive treatment of the primary with either curative intent radiotherapy and/or surgery
5. Patient has 1-5 sites of nodal or bony metastases on 68Ga-PSMA or 18F-DCFPyL PET/CT
6. Adequate haematological function as defined by:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count >150x 109/L
   * Haemoglobin ≥100 g/L
   * Creatinine Clearance ≥ 40mL/min (Cockcroft-Gault formula)
7. Assessed as suitable for SABR by a radiation oncologist
8. Patients must agree to use an adequate method of contraception
9. Have a performance status of 0-1 on the ECOG Performance Scale

Exclusion Criteria:

1. Prior systemic therapy for metastatic prostate cancer. Prior ADT is allowed but ADT within 6 months of screening for the study is not allowed. If patients have received prior ADT, serum testosterone levels must be above the lower limit of normal
2. Any visceral (AJCCC M1c) metastases
3. Symptomatic cord compression, or clinical or imaging findings concerning for impending cord compression
4. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
5. Has a known additional malignancy that is progressing or required active treatment in the last 2 years Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or carcinoma in situ such as breast cancer in situ that has undergone potentially curative therapy are not excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male aged 18 years or older at screening
Enrollment: 92 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the (bPFS) of SABR alone and SABR + 177Lu-PSMA | Through study completion, up until 12 months after the last patient commences treatment
  The biochemical progression free survival (bPFS) of SABR alone and SABR + 177Lu-prostate-specific membrane antigen (PSMA) in patients with oligometastatic prostate cancer undergoing PSMA positron emission tomography (PET) staging.

SECONDARY OUTCOMES:
The AEs according to CTCAE v5.0 | Through study completion, up until 4 months ± 10 days from the commencement of ADT following progression
  The type, grade and relationship to treatment of AEs will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0
The PSA-response rate | Through study completion, up until time of biochemical progression +/- 10 days
  PSA response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result
The ADT-free survival | Through study completion, up until biochemical progression +/- 10 days
  ADT-FS is defined as the time from randomisation to the date of initiation of androgen deprivation therapy or date of death due to any cause
The pattern of recurrence on PSMA PET | Time of biochemical progression +/-10 days
  Pattern of relapse will be evaluated on the PSMA PET at progression in relation to baseline PSMA PET, including: a) number of new sites of disease; b) location of new disease of disease (pelvic nodes, extra-pelvic nodes, bone, viscera); c) progression at prior sites (yes or no)
The patient reported quality of life | From the date of randomisation to the date of progression
  QoL will be assessed using the EORTC QLQC-30 and EQ-5D-5L questionnaires
The MDT PFS | Time point after Cycle 2 (28 days follow up post Cycle 2) until biochemical progression
  MDT PFS is defined as the time from first MDT after initial treatment to first documented subsequent disease progression (biochemical, or clinical using the same definition as the primary endpoint) or date of death, whichever comes first. Only patients who received MDT as the only treatment modality after initial treatment will be included.
The overall survival | Time point post randomisation to the date of death from any cause
  OS is defined as the time from randomisation to the date of death from any cause
Healthcare costs associated with delivering the intervention and management of AEs | Through study completion, an average of 3 years
  Health economic analysis is planned to assess the real-world cost-effectiveness and broader economic impact of using 177Lu-PSMA + SABR compared to SABR alone (if an effect is observed). Costs included in the analysis will focus on those relevant to the intervention (177Lu-PSMA) including treatment-related hospitalisations, clinic visits, PSMA PET scans, and associated medical service utilisation. Additionally, healthcare resource used and their associated costs including those associated with the complications arising from each study arm will be extracted from hospital administrative records and data collected during the trial (e.g., CTCAE v 5.0 Toxicity Record) and compared to provide an understanding of overall costs.
The PET-PFS | Through study completion, from the date of randomisation to the date of radiological progression or death from any cause, whichever comes first.
  PET-PFS is defined as the time from randomisation to the date of radiological progression on PSMA PET/CT scan or death due to any cause, whichever comes first. Patients alive without a rise in PSA will be censored at last PSA assessment

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof. Shankar Siva, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Dr Aravind S. Ravi Kumar, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (3):
- Australia (2):
  - Royal North Shore, St Leonards, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Sheba Medical Centre, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Individual requests for data sharing must be accompanied by ethical approval and will be considered at request